CLINICAL TRIAL: NCT00689273
Title: A 2-WEEK, RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL-GROUP, PHASE 2, MULTICENTER STUDY OF PF-04136309 IN SUBJECTS WITH OSTEOARTHRITIC PAIN OF THE KNEE
Brief Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study In Subjects With Osteoarthritic Pain Of The Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9421006
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
Keywords: PF-04136309 CCR2 osteoarthritic pain knee; phase 2 placebo multicenter double-blind placebo-controlled
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — PF-04136309

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-04136309 (Experimental)
  Interventions: Drug: PF-04136309
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04136309 — 125 mg capsules. Dose will be 4 capsules BID for 2 weeks for a total of 500 mg for each dosing interval.
  Arms: PF-04136309
Drug: Placebo — Placebo will be matched to PF-04136309. Dose, frequency, and duration same as PF-04136309.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety, tolerability, pharmacodynamics, and pharmacokinetics in patients with osteoarthritic pain of the knee. The most painful knee joint will be identified as the index joint at screening, and this joint will be used for all pain assessments throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, between the ages of 18 and 75 years inclusive
* Female subjects must be of non-childbearing potential and have a negative pregnancy test at Screening.
* Osteoarthritis of the knee of at least 6 months duration and meeting the American College of Rheumatology Criteria. For radiographic criteria the Xray must have been taken within the last 5 years. If none is available, one should be taken and the diagnostic criteria confirmed prior to randomization.
* Willing and able to discontinue all current analgesic therapy, including OTC pain medications and topical analgesics for OA pain, for period beginning with washout phase (lasting 2 days or 5 half-lives of patient's current analgesic medication prior to Day -6) and continuing for the entire duration of study. As an exception, acetaminophen may be used for non-joint related pain at doses ≤1 g/day at the discretion of a qualified member of the study team.
* If a subject has evidence or a history of clinically significant endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, renal, psychiatric, or neurological disease, the investigator must confirm that the disease is stable (at least 4 weeks) and under control.
* QTc interval ≤450 msec and a PR interval ≤210 msec on Screening ECG.

Exclusion Criteria:

* Pregnant or lactating females, and females of childbearing potential.
* Arthroscopy performed on index knee within 1 year of screening.
* Active depression as defined by or meeting The Hospital Anxiety and Depression Scale (HADS) of >10.
* Unwillingness to refrain from consumption of grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until completion of the study.
* First degree or higher AV block, defined as PR interval >210 msecs, bundle branch block, fascicular block or intraventricular conduction delay or clinically relevant abnormality on screening ECG.
* Active malignancy of any type or history of a malignancy within 10 years (with the exception of subjects with a history of treated basal cell carcinoma).
* Symptomatic OA of the hip ipsilateral to index knee which the patient considers more painful than the knee.
* Use of prohibited medications as listed below, in the absence of appropriate washout period. The following analgesic agents must be discontinued within 48 hours or 5 half lives of the analgesic being washed out prior to the baseline period (Day -6 to Day 0);

  * NSAIDs and selective COX-2 inhibitors;
  * Acetaminophen ( as an exception acetaminophen may be used for non-joint related pain at doses ≤1g/day);
  * Opioids.
  * Oral or I/M corticosteroids within 4 weeks prior to screening. I/A steroids within 12 weeks prior to baseline in study joint or any other joints within 4 weeks prior to baseline, or I/A hyaluronic acid within 24 weeks prior to baseline;
  * Use of concomitant medications that are CYP3A inhibitors or CYP3A inducers, or that are P-glycoprotein substrates within 48 hours or 5 half lives prior to baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2008-08-05 (Actual); Primary Completion 2008-11-27 (Actual); Study Completion 2008-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (18):
  - University Clinical Research-DeLand, LLC, DeLand, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Diagnostic Imaging Centers, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Covenant Health and Wellness Center, Chesterfield, Missouri
  - Metro Imaging St. Peters, City of Saint Peters, Missouri
  - Metro Imaging West County, Creve Coeur, Missouri
  - Analgesic Development Limited, New York, New York
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Statcare, Warwick, Rhode Island
  - Diagnostics Research Group, San Antonio, Texas
  - South Texas Radiology Group, San Antonio, Texas
  - Commonwealth Orthopaedics and Rehabilitation PC, Arlington, Virginia
  - IntegraTrials, LLC, Arlington, Virginia
  - United Hospital Center Clinical Trials Office, Clarksburg, West Virginia
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9421006&StudyName=Randomized%2C%20Double-Blind%2C%20Placebo-Controlled%2C%20Phase%202%20Study%20In%20Subjects%20%0AWith%20Osteoarthritic%20Pain%20Of%20The%20Knee

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04136309: Participants with osteoarthritis of knee received four 125 milligram (mg) capsules of PF-04136309, orally twice daily for 13 days and single morning dose on Day 14.
- Placebo: Participants with osteoarthritis of knee received placebo matched to four PF-04136309 125 mg capsules, orally twice daily for 13 days and single morning dose on Day 14.
Period: Overall Study
Arm/Group | PF-04136309 | Placebo
Started | 79 | 78
Treated | 78 | 78
Completed | 66 | 73
Not Completed | 13 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 3 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other | 6 | 2
Not completed — Randomized but not Treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04136309 | Placebo | Total
Number analyzed (Participants) | 78 | 78 | 156
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0
  18 to 44 years | 3 | 1 | 4
  45 to 64 years | 49 | 60 | 109
  Greater than or equal to 65 years | 26 | 17 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 37 | 37 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 33 | 31 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Domain Score at Week 2
Description: WOMAC: self-administered, disease-specific 24 item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness, and physical function in participants with osteoarthritis (OA) of the hip and/or knee. It consists of 3 domains: pain, stiffness and physical function. WOMAC pain domain consists of 5 questions scored on 5 point Likert scale (0=minimum pain to 4=maximum pain) where higher score indicates higher pain. It assesses amount of pain experienced due to OA in the study joint in past 48 hours. Total possible pain domain score calculated by addition of scores of each 5 questions ranged from: 0 (minimum) - 20 (maximum), higher scores indicate higher pain.
Time Frame: Baseline, Week 2
Population: FAS included all randomized participants who took at least 1 dose of study drug. Here 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 69 | 74
Units on a scale | -3.64 (0.41) | -3.15 (0.40)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Results were obtained from a mixed effect repeated measure model using unstructured covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect. One-sided alpha of 0.1 was used for the analysis; Test type: Superiority; p = 0.39, Mixed Models Analysis; Least Square (LS) Mean Difference = -0.49, 80% CI 2-sided [-1.23 to 0.24], Standard Error of Mean 0.57

2. Secondary Outcome: Change From Baseline in WOMAC Pain Domain Score at Week 1
Description: WOMAC: self-administered, disease-specific 24 item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness, and physical function in participants with OA of the hip and/or knee. It consists of 3 domains: pain, stiffness and physical function. WOMAC pain domain consists of 5 questions scored on 5 point Likert scale (0=minimum pain to 4=maximum pain) where higher score indicates higher pain. It assesses amount of pain experienced due to OA in the study joint in past 48 hours. Total possible pain domain score calculated by addition of scores of each 5 questions ranged from: 0 (minimum) - 20 (maximum), higher scores indicate higher pain.
Time Frame: Baseline, Week 1
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 76 | 76
Units on a scale | -2.74 (0.37) | -2.49 (0.37)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Results were obtained from a mixed effect repeated measure model using unstructured covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.63, Mixed Models Analysis; LS Mean Difference = -0.25, 80% CI 2-sided [-0.92 to 0.42], Standard Error of Mean 0.52

3. Secondary Outcome: Change From Baseline in WOMAC Stiffness Domain Score at Week 1 and Week 2
Description: WOMAC: self-administered, disease-specific 24 item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness, and physical function in participants with OA of the hip and/or knee. It consists of 3 domains: pain, stiffness and physical function. WOMAC stiffness domain consist of 2 questions scored on 5 point Likert scale (0=minimum stiffness to 4= maximum stiffness), higher score indicates higher stiffness. It assesses stiffness (sensation of decreased ease) due to OA in study joint in past 48 hours. Total possible stiffness domain score calculated by addition of scores of each 2 questions ranged from: 0 (minimum) to 8 (maximum), higher scores indicate higher stiffness.
Time Frame: Baseline, Weeks 1, 2
Population: FAS included all randomized participants who took at least 1 dose of study drug. Here, 'number analyzed' signifies participants evaluable for this outcome measure for specified time points.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 69 | 66
  Week 1 | -0.95 (0.19) | -0.78 (0.19)
  Week 2: number analyzed (Participants) | 62 | 63
  Week 2 | -1.39 (0.20) | -1.24 (0.20)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Week 1: Results were obtained from a mixed effect repeated measure model using unstructured covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.54, Mixed Models Analysis; LS Mean Difference = -0.17, 80% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; Week 2: Results were obtained from a mixed effect repeated measure model using unstructured covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.60, Mixed Models Analysis; LS Mean Difference = -0.15, 80% CI 2-sided [-0.51 to 0.21], Standard Error of Mean 0.28

4. Secondary Outcome: Change From Baseline in WOMAC Physical Function Domain Score at Week 1 and Week 2
Description: WOMAC: self-administered, disease-specific 24 item questionnaire which assesses clinically important, participant-relevant symptoms for pain, stiffness, and physical function in participants with OA of the hip and/or knee. It consists of 3 domains: pain, stiffness and physical function. WOMAC physical function consists of 17 questions scored on 5 point Likert scale (0=minimum physical impairment to 4=maximum physical impairment), higher score indicates worse function. It assesses worse function (ability to move/perform activity) due to OA in study joint in past 48 hours. Total possible score calculated by addition of scores of each 17 questions ranged from: 0 (minimum) to 68 (maximum), higher scores indicate worse function.
Time Frame: Baseline, Weeks 1, 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 69 | 66
  Week 1 | -8.63 (1.26) | -7.25 (1.29)
  Week 2: number analyzed (Participants) | 62 | 62
  Week 2 | -11.32 (1.41) | -8.90 (1.42)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.44, Mixed Models Analysis; LS Mean Difference = -1.38, 80% CI 2-sided [-3.69 to 0.94], Standard Error of Mean 1.80
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.23, Mixed Models Analysis; LS Mean Difference = -2.42, 80% CI 2-sided [-5.00 to 0.16], Standard Error of Mean 2.00

5. Secondary Outcome: Change From Baseline in WOMAC Total Score at Week 1 and Week 2
Description: WOMAC: self-administered, disease-specific instrument assessing clinically important, participant-relevant symptoms for pain, stiffness, physical function in participants with OA of the hip and/or knee. Index consists of 24 questions: 5 (pain), 2 (stiffness), 17 (physical function). Each question was assessed on a 5-point Likert scale (0= none to 4=extreme), higher score indicates worse function. Total WOMAC Score: summation of 24 component item scores, without any correction for relative importance of different subscales. Total score range 0 (minimum) to 96 (maximum), higher score indicate higher symptoms.
Time Frame: Baseline, Weeks 1, 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 69 | 66
  Week 1 | -12.31 (1.72) | -10.54 (1.76)
  Week 2: number analyzed (Participants) | 62 | 62
  Week 2 | -16.24 (1.96) | -13.22 (1.98)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.48, Mixed Models Analysis; LS Mean Difference = -1.76, 80% CI 2-sided [-4.94 to 1.41], Standard Error of Mean 2.46
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.28, Mixed Models Analysis; LS Mean Difference = -3.02, 80% CI 2-sided [-6.61 to 0.57], Standard Error of Mean 2.79

6. Secondary Outcome: Change From Baseline in WOMAC Importance Weighted Total Score at Week 1 and Week 2
Description: WOMAC: self-administered, disease-specific instrument assessing clinically important, participant-relevant symptoms for pain, stiffness, physical function in participants with OA of hip or knee. Index consists of 24 questions: 5 (pain), 2 (stiffness), 17 (physical function). Each question was assessed on a 5-point Likert scale; score range: 0 (none) to 4 (extreme) where higher score indicates worse function. Importance-weighted total WOMAC score weighs 3 subscales of pain, stiffness, physical function using factors of 0.42, 0.21, and 0.37 to account for relative importance. Total score calculated by applying factors and summing all domains ranged from 0 (minimum) to 35.24 (maximum), higher score indicate higher symptoms.
Time Frame: Baseline, Weeks 1, 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 69 | 66
  Week 1 | -4.54 (0.63) | -3.90 (0.65)
  Week 2: number analyzed (Participants) | 62 | 62
  Week 2 | -5.97 (0.72) | -4.84 (0.73)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.48, Mixed Models Analysis; LS Mean Difference = -0.65, 80% CI 2-sided [-1.81 to 0.52], Standard Error of Mean 0.91
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.28, Mixed Models Analysis; LS Mean Difference = -1.12, 80% CI 2-sided [-2.45 to 0.20], Standard Error of Mean 1.03

7. Secondary Outcome: Change From Baseline in 11 Point Numeric Pain Rating Scale (NRS) at Week 1 and Week 2 (Weekly Average)
Description: NRS: participant rated their daily pain on 11-point Likert scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain.
Time Frame: Baseline, Weeks 1, 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 77 | 78
  Week 1 | -0.83 (0.14) | -0.62 (0.14)
  Week 2: number analyzed (Participants) | 72 | 75
  Week 2 | -1.56 (0.20) | -1.14 (0.20)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.28, Mixed Models Analysis; LS Mean Difference = -0.21, 80% CI 2-sided [-0.46 to 0.04], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.14, Mixed Models Analysis; LS Mean Difference = -0.42, 80% CI 2-sided [-0.78 to -0.06], Standard Error of Mean 0.28

8. Secondary Outcome: Change From Baseline in 11 Point NRS at Each Day From Day 1 to Day 14
Description: as for outcome 7
Time Frame: Baseline, Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Day 1: number analyzed (Participants) | 76 | 78
  Day 1 | -0.26 (0.20) | -0.09 (0.19)
  Day 2: number analyzed (Participants) | 74 | 76
  Day 2 | -0.67 (0.20) | -0.22 (0.20)
  Day 3: number analyzed (Participants) | 77 | 76
  Day 3 | -0.81 (0.20) | -0.46 (0.20)
  Day 4: number analyzed (Participants) | 73 | 76
  Day 4 | -0.91 (0.20) | -0.58 (0.20)
  Day 5: number analyzed (Participants) | 76 | 75
  Day 5 | -1.02 (0.20) | -0.80 (0.20)
  Day 6: number analyzed (Participants) | 75 | 76
  Day 6 | -1.11 (0.20) | -0.97 (0.20)
  Day 7: number analyzed (Participants) | 72 | 77
  Day 7 | -1.23 (0.20) | -1.04 (0.19)
  Day 8: number analyzed (Participants) | 72 | 73
  Day 8 | -1.50 (0.20) | -1.04 (0.20)
  Day 9: number analyzed (Participants) | 70 | 74
  Day 9 | -1.35 (0.20) | -1.03 (0.20)
  Day 10: number analyzed (Participants) | 69 | 72
  Day 10 | -1.49 (0.20) | -0.84 (0.20)
  Day 11: number analyzed (Participants) | 69 | 73
  Day 11 | -1.60 (0.20) | -1.03 (0.20)
  Day 12: number analyzed (Participants) | 68 | 71
  Day 12 | -1.82 (0.20) | -1.23 (0.20)
  Day 13: number analyzed (Participants) | 66 | 72
  Day 13 | -1.76 (0.20) | -1.43 (0.20)
  Day 14: number analyzed (Participants) | 67 | 68
  Day 14 | -1.82 (0.20) | -1.36 (0.20)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Day 1: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.55, Mixed Models Analysis; LS Mean Difference = -0.17, 80% CI 2-sided [-0.52 to 0.19], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; Day 2: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.11, Mixed Models Analysis; LS Mean Difference = -0.45, 80% CI 2-sided [-0.81 to -0.09], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: PF-04136309 vs Placebo; Day 3: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.20, Mixed Models Analysis; LS Mean Difference = -0.35, 80% CI 2-sided [-0.71 to 0.00], Standard Error of Mean 0.28
Statistical Analysis 4: Comparison: PF-04136309 vs Placebo; Day 4: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.23, Mixed Models Analysis; LS Mean Difference = -0.33, 80% CI 2-sided [-0.69 to 0.02], Standard Error of Mean 0.28
Statistical Analysis 5: Comparison: PF-04136309 vs Placebo; Day 5: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.41, Mixed Models Analysis; LS Mean Difference = -0.23, 80% CI 2-sided [-0.58 to 0.13], Standard Deviation 0.28
Statistical Analysis 6: Comparison: PF-04136309 vs Placebo; Day 6: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.62, Mixed Models Analysis; LS Mean Difference = -0.14, 80% CI 2-sided [-0.49 to 0.22], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: PF-04136309 vs Placebo; Day 7: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.49, Mixed Models Analysis; LS Mean Difference = -0.19, 80% CI 2-sided [-0.55 to 0.16], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: PF-04136309 vs Placebo; Day 8: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.10, Mixed Models Analysis; LS Mean Difference = -0.46, 80% CI 2-sided [-0.81 to -0.10], Standard Deviation 0.28
Statistical Analysis 9: Comparison: PF-04136309 vs Placebo; Day 9: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.24, Mixed Models Analysis; LS Mean Difference = -0.33, 80% CI 2-sided [-0.69 to 0.03], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: PF-04136309 vs Placebo; Day 10: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.02, Mixed Models Analysis; LS Mean Difference = -0.65, 80% CI 2-sided [-1.01 to -0.28], Standard Error of Mean 0.28
Statistical Analysis 11: Comparison: PF-04136309 vs Placebo; Day 11: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.04, Mixed Models Analysis; LS Mean Difference = -0.57, 80% CI 2-sided [-0.93 to -0.21], Standard Error of Mean 0.28
Statistical Analysis 12: Comparison: PF-04136309 vs Placebo; Day 12: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.04, Mixed Models Analysis; LS Mean Difference = -0.59, 80% CI 2-sided [-0.95 to -0.23], Standard Error of Mean 0.28
Statistical Analysis 13: Comparison: PF-04136309 vs Placebo; Day 13: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.24, Mixed Models Analysis; LS Mean Difference = -0.33, 80% CI 2-sided [-0.70 to 0.03], Standard Error of Mean 0.28
Statistical Analysis 14: Comparison: PF-04136309 vs Placebo; Day 14: Results were obtained from a mixed effect repeated measure model using compound symmetry covariance matrix. The model included random-effect terms for participant, and fixed-effect terms for baseline response, treatment group, time, treatment-by-time interaction, and country effect; Test type: Superiority; p = 0.11, Mixed Models Analysis; Slope = -0.45, 80% CI 2-sided [-0.82 to -0.09], Standard Error of Mean 0.28

9. Secondary Outcome: Number of Participants With at Least a 30 Percent (%) and 50% Reduction in Average Weekly Pain Score at Week 2: Last Observation Carried Forward (LOCF)
Description: Participant rated their daily pain on 11-point Likert scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain. In this outcome measure number of participants with at least 30% and 50% reduction in average weekly pain score at Week 2 from Baseline are reported. Average weekly score at Week 2 was average of daily pain scores from Day 8 to Day 14 and at Baseline it was average of daily pain scores from Day -6 to Day 0.
Time Frame: Baseline, Week 2
Population: FAS included all randomized participants who took at least 1 dose of study drug. LOCF method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  30% Reduction | 27 | 20
  50% Reduction | 14 | 10
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; 30% Reduction; Test type: Superiority; p = 0.22, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; 50% Reduction; Test type: Superiority; p = 0.38, Cochran-Mantel-Haenszel

10. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritic Condition at Week 1 and Week 2
Description: Participants answered the following question: "Considering all the ways your arthritis affects you, how are you doing today?" Participants rated their condition using the scale assessing the symptoms and limitations to carry out normal daily activities. Score ranged from 1 to 5; where 1= very good (No symptoms and limitations); 2= good (mild symptoms and no limitations); 3= fair (moderate symptoms and some limitations); 4= poor (severe symptoms and inability to carry out most activities); and 5= very Poor (very severe, intolerable symptoms and inability to carry out all activities). Higher scores indicated more limitations in carrying out normal activities.
Time Frame: Baseline, Weeks 1, 2
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Units on a scale
  Week 1: number analyzed (Participants) | 69 | 66
  Week 1 | -0.42 (0.09) | -0.32 (0.09)
  Week 2: number analyzed (Participants) | 62 | 63
  Week 2 | -0.56 (0.09) | -0.44 (0.09)
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.45, Mixed Models Analysis; LS Mean Difference = -0.10, 80% CI 2-sided [-0.27 to 0.07], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.37, Mixed Models Analysis; LS Mean Difference = -0.12, 80% CI 2-sided [-0.29 to 0.05], Standard Error of Mean 0.13

11. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. SAE was defined as any untoward medical occurrence at any dose that: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Treatment emergent AEs included both SAEs and all non-SAEs.
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  Treatment Emergent AEs | 22 | 21
  Treatment Emergent SAEs | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment Related AEs and SAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Treatment emergent AEs included both SAEs and all non-SAEs. A treatment-related SAE was a treatment-related AE and was defined as any untoward medical occurrence at any dose that: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. Relatedness to study drug was assessed by the investigator.
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  Treatment Emergent Treatment Related AEs | 13 | 16
  Treatment Emergent Treatment Related SAEs | 0 | 0

13. Other Pre Specified Outcome: Number of Participants Who Discontinued Due to Treatment Emergent AEs and Treatment Emergent Treatment Related AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug.
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  Treatment Emergent AEs | 3 | 1
  Treatment Emergent Treatment Related AEs | 1 | 1

14. Other Pre Specified Outcome: Number of Treatment-Emergent AEs by Severity
Description: Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. The severity grades (mild, moderate and severe) were defined as - Mild: did not interfere with participant's usual function, Moderate: Interfered to some extent with participant's usual function and Severe: Interfered significantly with participant's usual function.
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Events
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Events
  Mild | 24 | 29
  Moderate | 2 | 9
  Severe | 2 | 1

15. Other Pre Specified Outcome: Number of Treatment-Emergent Treatment-Related AEs by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Treatment-emergent AEs were events that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. The severity grades (mild, moderate and severe) were defined as - Mild: did not interfere with participant's usual function, Moderate: Interfered to some extent with participant's usual function and Severe: Interfered significantly with participant's usual function.
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Events
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Events
  Mild | 13 | 18
  Moderate | 1 | 4
  Severe | 1 | 1

16. Other Pre Specified Outcome: Number of Participants Who Discontinued Due to Treatment-Emergent AEs According to Severity
Description: as for outcome 14
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants
  Mild | 1 | 1
  Moderate | 1 | 0
  Severe | 1 | 0

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Blood Pressure and Pulse Rate
Description: Criteria for clinical significance: sitting, standing or supine pulse rate <40 beats per minute (bpm) or >120 bpm; sitting, standing or supine diastolic blood pressure < 50 millimeter of mercury (mmHg); sitting, standing or supine systolic blood pressure < 90 mmHg. Clinical significance was judged by the investigator.
Time Frame: From Baseline up to Week 2
Population: FAS included all randomized participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 78 | 78
Participants | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Change (Increase) From Baseline in Electrocardiogram (ECG) Parameters
Description: Change (increase) from baseline of greater than or equal to (>=) 25% in maximum PR Interval and maximum QRS complex in milliseconds (msec). Change (increase) from baseline of >= 30 msec and less than (<) 60 msec or change >= 60 msec in maximum QTc and maximum QT interval with Fridericia's Correction (QTcF).
Time Frame: Baseline up to Week 2
Population: FAS included all randomized participants who took at least 1 dose of study drug. Here 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. Here, 'number analyzed' signifies participants evaluable for this outcome measure for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 77 | 77
Participants
  Maximum PR Interval increase from baseline; change >=25% | 0 | 0
  Maximum QRS Complex increase from baseline; change >=25% | 0 | 0
  Maximum QTc Interval increase from baseline; Change >=30 msec and < 60 msec: number analyzed (Participants) | 76 | 77
  Maximum QTc Interval increase from baseline; Change >=30 msec and < 60 msec | 1 | 0
  Maximum QTc Interval increase from baseline; Change >=60 msec: number analyzed (Participants) | 76 | 77
  Maximum QTc Interval increase from baseline; Change >=60 msec | 1 | 0
  Maximum QTcF Interval increase from baseline; Change >=30 msec and < 60 msec | 1 | 0
  Maximum QTcF Interval increase from baseline; Change >=60 msec | 1 | 0

19. Other Pre Specified Outcome: Plasma Concentration Versus Time of PF-04136309
Description: In this outcome measure data for reporting arm PF-04136309 was collected and reported as planned.
Time Frame: Day 1 and Day 14: Pre-dose and 6,7 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04136309
Number analyzed (Participants) | 78
Nanogram per milliliter
  Day 1: pre-dose: number analyzed (Participants) | 56
  Day 1: pre-dose | 257.90 (276.38)
  Day 1: 6 hours post-dose: number analyzed (Participants) | 14
  Day 1: 6 hours post-dose | 587.54 (626.53)
  Day 1: 7 hours post-dose: number analyzed (Participants) | 12
  Day 1: 7 hours post-dose | 590.85 (615.06)
  Day 14: 0 hours pre-dose: number analyzed (Participants) | 63
  Day 14: 0 hours pre-dose | 227.42 (259.21)
  Day 14: 6 hours post-dose: number analyzed (Participants) | 6
  Day 14: 6 hours post-dose | 388.00 (244.98)
  Day 14: 7 hours post-dose: number analyzed (Participants) | 7
  Day 14: 7 hours post-dose | 426.14 (266.11)

20. Other Pre Specified Outcome: Change From Baseline in Absolute Monocyte Count at Day 14
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Thousand cells per millimeter cube
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 77 | 77
Thousand cells per millimeter cube | -0.13 [-0.19 to -0.04] | -0.01 [-0.06 to 0.06]

21. Other Pre Specified Outcome: Change From Baseline in Percent Monocytes at Day 14
Description: Monocytes (percent) were derived as monocyte absolute counts per white blood cell absolute counts*100.
Time Frame: Baseline, Day 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent monocytes
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 77 | 77
Percent monocytes | -1.7 [-2.7 to -0.1] | 0.0 [-0.8 to 1.0]

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after last dose of study drug (up to Day 44)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study. FAS included all randomized participants who received at least 1 dose of study drug.
Arm/Group | PF-04136309 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/78
Other Adverse Events (participants affected / at risk) | 22/78 | 21/78
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04136309 (N=78) | Placebo (N=78)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Ulcer (General disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Blood glucose increased (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 6 | 3
Somnolence (Nervous system disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.